CLINICAL TRIAL: NCT05434611
Title: Role of Calcium Binding Protein S100A12 in Diagnosis and Prognosis of Kawasaki Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Yangtze University (Other)
Responsible Party: Principal Investigator, Pan Yan, Attending physician, The First Affiliated Hospital of Yangtze University
Other Study IDs: PYan
Record Dates: First submitted 2022-06-16; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Diagnoses Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kawasaki disease: All children with Kawasaki disease met the diagnostic criteria for Kawasaki disease revised by the American Heart Association in 2017.
  Interventions: Diagnostic Test: S100A12
- Healthy controls: Healthy control group were healthy children who underwent outpatient physical examination.
  Interventions: Diagnostic Test: S100A12

INTERVENTIONS:
Diagnostic Test: S100A12 — The early dynamic detection of S100A12 was used to determine whether it was an auxiliary diagnostic index for Kawasaki disease

SUMMARY:
Recent studies showed that the value of c100A12 increased in children with Kawasaki disease, and decreased rapidly after treatment with gamma globulin. In kawasaki disease with coronary artery dilatation, S100A12 levels are elevated in the acute phase of Kawasaki disease and continue for some time in the convalescence phase before gradually decreasing. However, the number of patients included in previous studies was small and the follow-up time was short. In this study, 100 children with Kawasaki disease who were admitted to Wuhan Children's Hospital, Jingzhou First People's Hospital and Renhe Hospital affiliated to China Three Gorges University from December 2021 to December 2023 were selected as the research objects, and 100 children with healthy physical examination were selected as the control group during the same period. To investigate whether S100A12 increased significantly in the acute phase of Kawasaki disease compared with a healthy control group. To study whether S100A12 value increased rather than decreased in kawasaki disease that did not respond to gamma globulin treatment after gamma globulin treatment. At the same time, to study whether the increase of S100A12 in kawasaki disease convalescence indicates coronary aneurysm.

DETAILED DESCRIPTION:
S100A12 was determined using the ELISA kit and according to the instructions.

ELIGIBILITY:
Inclusion Criteria:

▪Diagnostic criteria of Kawasaki disease revised by the American Heart Association in 2017

Exclusion Criteria:

* Scarlet fever
* Drug allergy syndrome
* Stevens-Johnson syndrome
* Toxic shock syndrome
* Adenovirus infection
* Epstein-Barr(EB) virus infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The case group consisted of 50 hospitalized children with Kawasaki disease. The healthy control group consisted of 50 healthy children.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
S100A12 | From date of randomization until the date of first documented progression, whichever came first, assessed up to 18 months
  S100A12 was increased in children with Kawasaki disease and decreased after gamma globulin treatment

SECONDARY OUTCOMES:
CRP | From date of randomization until the date of first documented progression, whichever came first, assessed up to 18 months
  Measure the CRP value

CONTACTS AND LOCATIONS:
Overall Officials: Qihong Fan, Dr., Principal Investigator — Yangtze University

IPD SHARING:
Plan to Share IPD: No